CLINICAL TRIAL: NCT06119022
Title: CT Myocardial Perfusion Imaging to Guide the Diagnosis and Treatment of Patients With Stable Coronary Artery Disease: a Randomized Controlled Study (POTENTIAL)
Brief Title: CT Myocardial Perfusion to Guide the Diagnosis and Treatment of Patients With Stable Coronary Artery Disease (POTENTIAL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Bin Lu, Director of Radiologic Imaging, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-GSP-GG-21
Record Dates: First submitted 2023-10-22; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Treatment Decision, Coronary Artery Disease
Keywords: CT myocardial perfusion imaging; Coronary artery disease; clinical pathway; SPECT myocardial perfusion imaging
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CT-MPI guided without myocardial ischemia (Experimental): There was no evidence of myocardial ischemia in patients with coronary heart disease by CT-MPI
  Interventions: Other: routine medical treatment
- CT-MPI guided with myocardial ischemia (Experimental): There was positive evidence of myocardial ischemia in patients with coronary heart disease by CT-MPI
  Interventions: Procedure: Invasive coronary angiography
- SPECT-MPI guided without myocardial ischemia (Active Comparator): There was no evidence of myocardial ischemia in patients with coronary heart disease by SPECT-MPI
  Interventions: Other: routine medical treatment
- SPECT-MPI guided with myocardial ischemia (Active Comparator): There was positive evidence of myocardial ischemia in patients with coronary heart disease by SPECT-MPI
  Interventions: Procedure: Invasive coronary angiography

INTERVENTIONS:
Procedure: Invasive coronary angiography — Patients with positive myocardial ischemia either in CT-MPI guided arm or SPECT-MPI guided arm will scheduled to undergo invasive coronary angiography.
  Arms: CT-MPI guided with myocardial ischemia; SPECT-MPI guided with myocardial ischemia
Other: routine medical treatment — Patients with negative myocardial ischemia either in CT-MPI guided arm or SPECT-MPI guided arm will scheduled to have routine medical therapy instead of invasive coronary angiography.
  Arms: CT-MPI guided without myocardial ischemia; SPECT-MPI guided without myocardial ischemia

SUMMARY:
The overall goal of this project is to compare the non-revascularization rate of coronary angiography in patients with stable coronary artery disease (CAD) within 90 days after CT myocardial perfusion imaging (CT-MPI) or Single-Photon Emission Computed Tomography myocardial perfusion imaging (SPECT-MPI), and 1-year major adverse cardiovascular events (MACE).

DETAILED DESCRIPTION:
Participants will be patients with proven coronary artery disease (CAD) who are scheduled randomized to undergo CT Myocardial Perfusion Imaging (CT-MPI) or Single-Photon Emission Computed Tomography myocardial perfusion imaging (SPECT-MPI) to evaluate myocardium ischemia. Those patients with positive myocardial ischemia will scheduled to undergo invasive coronary angiography (ICA), and those without myocardial ischemia will have optical medical therapy. The purpose of the study is to verify that CT-MPI guided clinical pathways are not inferior to SPECT-MPI pathways in downstream treatment decision making and safety assessment. In order to achieve this aim, the study team will compare the non-revascularization rate of ICA within 90 days after CT-MPI and SPECT-MPI. 1-year major adverse cardiovascular events (MACE) will be also compared.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with stable chest pain who have undergone coronary CT angiography and have 50-90% stenosis in at least one vessel > 2mm in diameter
* Able to provide signed informed consent

Exclusion Criteria:

* Suspected or confirmed acute coronary syndrome
* Evidence of clinical instability or need for an emergent procedure
* History of percutaneous coronary stent implantation, history of coronary artery bypass grafting, or history of myocardial infarction
* Left main artery stenosis ≥ 50%
* Severe heart failure (New York Heart Association (NYHA) ≥III)
* Estimated glomerular filtration rate < 60 mL/min/1.73 m2
* Contraindicated to use contrast agents, beta-blockers, nitrates or adenosine drugs
* Acute episodes of bronchial asthma or chronic obstructive pulmonary disease
* II or III degree atrioventricular block
* History of pacemaker or implantable cardioverter defibrillator implantation
* Combined with other cardiovascular diseases including cardiomyopathy, congenital heart disease, valvular heart disease, pulmonary vascular disease, pericardial disease, etc
* Pregnant or trying to be pregnant
* Combined with any other serious disease, life expectancy <1 year
* Any condition leading to possible inability to comply with the protocol procedures and follow-up
* Currently participating in any other clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of non-revascularization treatment of the two arms | within 90 days after CT-MPI or SPECT-MPI examination
  The incidence of conventional angiography not leading to revascularization within 90 days after CT-MPI or SPECT-MPI.

SECONDARY OUTCOMES:
The rate of major adverse cardiovascular events of the two arms | One year after CT-MPI or SPECT-MPI
  The composition of all-cause death, non-fatal myocardial infarction, stroke, revascularization, and hospital admissions for unstable angina.
Difference in quality of Life of the two arms | One year after CT-MPI or SPECT-MPI
  The Seattle Angina Questionnaire
Difference in cost of the two arms | One year after CT-MPI or SPECT-MPI
  Total clinical cost
Difference in cumulative radiation exposure dose of the two arms | Total cumulative radiation exposure dose during CT-MPI or SPECT-MPI and invasive coronary angiography within one year
  Total cumulative radiation exposure dose

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Fu Wai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - The First Affiliated Hosptial of Zhengzhou University, Zhengzhou, Henan
  - The Second Norman Bethune Hospital of Jilin University, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No